CLINICAL TRIAL: NCT07406100
Title: A Pilot Investigation of the Competence in Romance and Understanding Sexual Health Curriculum
Brief Title: Piloting the Competence in Romance and Understanding Sexual Health Curriculum
Acronym: CRUSH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Susan Faja, Associate Professor, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: FP01037275; 2009 (Other Grant/Funding Number: Organization for Autism Research)
Record Dates: First submitted 2026-01-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Autism; Autism Disorder; Autism Spectrum Disorder
Keywords: sexual health; romantic relationships
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Mental Competency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRUSH Intervention (Experimental): Participants will receive the CRUSH Curriculum
  Interventions: Behavioral: Competence in Romance and Understanding Sexual Health (CRUSH)
- Waitlist (No Intervention): Will be invited to receive the CRUSH intervention at the end of the study period

INTERVENTIONS:
Behavioral: Competence in Romance and Understanding Sexual Health (CRUSH) — Manualized curriculum targeting sexual health and behavior in intimate relationships designed to meet the specific needs of autistic adults
  Arms: CRUSH Intervention

SUMMARY:
The goal of this clinical trial is to learn whether the CRUSH curriculum is possible (feasible), whether it fits the needs of the adults it is designed for (acceptable), and shows initial signs of being helpful (efficacious). CRUSH is a group-based behavioral intervention plus 1-1 coaching designed to provide sexual education and improve the skills of autistic adults for intimate relationships.

The main goals of the project are to:

* Evaluate the feasibility and acceptability of the CRUSH curriculum in the context of a clinical trial with a waitlist control condition.
* Initial exploration of how the CRUSH curriculum works and whether it is helpful.

Participants will complete:

* A screening call.
* Confirmation of clinical characteristics (autism features, language ability, cognitive ability).
* 3 visits to assess knowledge and behaviors related to dating and sexual health at each point throughout the training curriculum (before beginning, midway, and after finishing).
* 20 sessions of the CRUSH curriculum plus 1-1 coaching sessions. After each session, provide feedback about the session.

DETAILED DESCRIPTION:
There are currently no evidence-based interventions to improve the dating and sexual health of autistic adults. The CRUSH (Competence in Romance and Understanding Sexual Health) Curriculum was designed to address this critical gap, which was piloted with a small group of participants. This study is a pilot program of the CRUSH curriculum for 40 participants to acquire initial feasibility and acceptability data. It will also test the feasibility and acceptability of the measurement battery for potential inclusion in future clinical trials. The goal of this clinical trial is to learn whether the CRUSH curriculum is possible (feasible), whether it fits the needs of the adults it is designed for (acceptable), how it works (mechanism), and shows initial signs of being helpful (efficacious). CRUSH is a group-based behavioral intervention plus 1-1 coaching designed to provide sexual education and improve the skills of autistic adults for intimate relationships.

The main goals of the project are to:

* Evaluate the feasibility and acceptability of the CRUSH curriculum in the context of a clinical trial with a waitlist control condition.
* Initial exploration of how the CRUSH curriculum works and whether it is helpful.

Participants will complete:

* A screening call.
* Confirmation of clinical characteristics (autism features, language ability, cognitive ability).
* 3 visits to assess knowledge and behaviors related to dating and sexual health at each point throughout the training curriculum (before beginning, midway, and after finishing).
* 20 sessions of the CRUSH curriculum plus 1-1 coaching sessions. After each session, provide feedback about the session.

ELIGIBILITY:
Inclusion Criteria:

* 18;0 to 30;11 years old;
* Either documentation of a prior diagnosis of autism spectrum disorder or receipt of services based on an autism spectrum diagnosis OR self identification as being autistic / on the autism spectrum and meeting the clinical cut-off on either the Autism Diagnostic Observation Schedule or the Autism Spectrum Quotient;
* Ability to provide consent for the protocol and understand task demands. The Wechsler Abbreviated Scale of Intelligence, Second Edition (WASI-2) may be used to confirm cognitive level. In prior work, adults with full scale IQ of 70 or above on the WASI-2 typically meet this criterion, but a licensed clinician will review individuals who fall below an IQ of 70 on an individual basis to determine eligibility;
* Fluent in English.

Exclusion Criteria:

* Non-English-speaking participants (less than 50% of speech in English);
* Known genetic etiology of ASD (e.g., Fragile X);
* Major mental illness (e.g., bipolar disorder, schizophrenia, or psychosis);
* Medical conditions that impact sexual function (e.g., pituitary tumor);
* Significant sensory, motor, or physical conditions that would prevent valid participation in assessments or intervention;
* Live more than 50 miles from the site in Brookline, MA where intervention and assessment sessions will be offered.
* Receipt of other sexual health/dating curricula as an adult.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability Rating Scale | Within one day of each intervention session and at the Baseline, Midpoint (10 weeks), and Post-intervention visit (20 weeks)
  This is the primary acceptability outcome. Likert ratings with a 5-pt scale
Sexual Vocabulary Test - Pragmatics Total Score | At the Baseline, Midpoint (10-weeks), and Post-intervention (20-weeks) visits
  This is the primary measure of target engagement. A measure of the ability to provide definitions of sexual health terms to be used as a measure of target engagement - the primary dependent variable measures pragmatic language (e.g., slang) when discussing sexual health terms. Accuracy (knowledge of sexual health terms) is also collected as a secondary variable.
Psychosexual Knowledge Test | At the Baseline, Midpoint (10-weeks), and Post-intervention (20-weeks) visits
  This is the primary clinical outcome measure and assesses changes in the information participants have. This task was adapted for the first RCT of a sexual health curriculum developed for autistic adolescents to assess changes in information. It includes 35 multiple choice and 2 open-ended items that are scored as correct or incorrect.

SECONDARY OUTCOMES:
Feasibility Assessment | Within one day of each intervention session and at the Baseline, Midpoint (10 weeks), and Post-intervention visit (20 weeks)
  Attrition rates; Missing data rates for assessment instruments

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Two Brookline Place, Brookline, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No